CLINICAL TRIAL: NCT01945567
Title: Randomised Crossover Trial of Deep Brain Stimulation of Differential Posterior Subthalamic Area Regions in Parkinson's Disease and Tremor
Brief Title: Randomised Crossover Trial of DBS of Differential PSA Regions in Parkinson's Disease and Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Responsible Party: Principal Investigator, Professor Christopher Lind, Professor, School of Surgery, The University of Western Australia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-039
Record Dates: First submitted 2013-09-14; First posted 2013-09-18 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Parkinson's Disease; Tremor
Keywords: Parkinson's disease; Essential tremor; Tremor; Deep brain stimulation; Posterior subthalamic area; Zona incerta
MeSH Terms: conditions — Parkinson Disease; Tremor; Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dorsal zona incerta (Experimental): Up to 3 mA, 60 us, 130 Hz deep brain stimulation
  Interventions: Device: Up to 3 mA, 60 us, 130 Hz deep brain stimulation
- Caudal zona incerta (Experimental): Up to 3 mA, 60 us, 130 Hz deep brain stimulation
  Interventions: Device: Up to 3 mA, 60 us, 130 Hz deep brain stimulation
- Empirical deep brain stimulation (Experimental): Empirical unblinded deep brain stimulation programming using any posterior subthalamic area electrode contact(s) and stimulation parameters to optimise clinical outcome.
  Interventions: Device: Empirical unblinded deep brain stimulation programming

INTERVENTIONS:
Device: Up to 3 mA, 60 us, 130 Hz deep brain stimulation
  Arms: Caudal zona incerta; Dorsal zona incerta
Device: Empirical unblinded deep brain stimulation programming
  Arms: Empirical deep brain stimulation

SUMMARY:
The posterior subthalamic area holds promise as a target region for deep brain stimulation in tremor and Parkinson's disease. Using the magnetic resonance-directed implantable guide tube surgical technique, subregions of the posterior subthalamic area can be individually targetted on a single electrode lead trajectory. The hypothesis is that the caudal zona incerta may provide improved control of movement disorder symptoms than the more commonly stimulated dorsal zona incerta.

DETAILED DESCRIPTION:
Randomisation between two treatment locations each programmed up to 3 milliamps in amplitude for 3 months: (1) caudal zona incerta and (2) dorsal zona incerta. This 6-month-long randomised phase is followed by 6 months of unblinded individualised empirically optimised settings programmed by a neurologist. Each of the three treatment periods ends with a full clinical, functional and quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

* Medication-refractory tremor and/or Parkinson's disease as defined by UK Brain Bank criteria with either inadequate control of motor fluctuations or dyskinesia despite optimised medical therapy

Exclusion Criteria:

* Significant cognitive, psychiatric and medical co-morbidities
* Dementia with mini mental state examination score of less than 25/30
* Limited life expectancy due to a co-morbid condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline United Parkinsons Disease Rating Scale Part III at 3 months | 3 months
  At end of first randomised crossover trial period
Change from baseline United Parkinsons Disease Rating Scale Part III at 6 months | 6 months
  At end of second randomised crossover trial period
Change from baseline United Parkinsons Disease Rating Scale Part III at 12 months | 12 months
  At end of non-randomised empirical deep brain stimulator programming period
Change from baseline Fahn Tolosa Marin tremor scale at 3 months | 3 months
  At end of first randomised crossover trial period for tremor patients
Change from baseline Fahn Tolosa Marin tremor scale at 6 months | 6 months
  At end of second randomised crossover trial period for tremor patients
Change from baseline Fahn Tolosa Marin tremor scale at 12 months | 12 months
  At end of empirical deep brain stimulator programming period for tremor patients

SECONDARY OUTCOMES:
Change from baseline ON-OFF diary at 3 months | 3 months
  For Parkinson's disease
Change from baseline ON-OFF diary at 6 months | 6 months
  For Parkinson's disease
Change from baseline ON-OFF diary at 12 months | 12 months
  For Parkinson's disease
Adverse events | 12 months
  Any adverse medical event from date of randomization until the date of first documented adverse event or date of death from any cause, whichever came first, assessed up to 12 months
Change from baseline Short form 36 at 3 months | 3 months
  At end of first randomised crossover period
Change from baseline Short form 36 at 6 months | 6 months
  At end of second randomised crossover period
Change from baseline Short form 36 at 12 months | 12 months
  At end of empirical deep brain stimulator programming period
Change from baseline Parkinsons Disease Quality of Life 39 at 3 months | 3 months
  At end of first randomised crossover period for Parkinsons disease
Change from baseline Parkinsons Disease Quality of Life 39 at 6 months | 6 months
  At end of second randomised crossover period for Parkinsons disease
Change from baseline Parkinsons Disease Quality of Life 39 at 12 months | 12 months
  At end of empirical deep brain stimulator programming period for Parkinsons disease
Change from baseline L-dopa equivalent dose at 3 months | 3 months
  At end of first randomised crossover period for Parkinsons disease
Change from baseline L-dopa equivalent dose at 6 months | 3 months
  At end of second randomised crossover period for Parkinsons disease
Change from baseline L-dopa equivalent dose at 12 months | 12 months
  At end of empirical deep brain stimulator programming period for Parkinsons disease
Change from baseline neuropsychological battery at 3 months | 3 months
  At end of first randomised crossover period
Change from baseline neuropsychological battery at 6 months | 6 months
  At end of second randomised crossover period
Change from baseline neuropsychological battery at 12 months | 12 months
  At end of empirical deep brain stimulator programming period
Change from baseline verbal fluency at 3 months | 3 months
  At end of first randomised crossover period
Change from baseline verbal fluency at 6 months | 6 months
  At end of second randomised crossover period
Change from baseline verbal fluency at 12 months | 12 months
  At end of empirical deep brain stimulator programming period
Change from baseline Mini-International Neuropsychiatric Interview Plus at 3 months | 3 months
  At end of first randomised crossover period
Change from baseline Mini-International Neuropsychiatric Interview Plus at 6 months | 6 months
  At end of second randomised crossover period
Change from baseline Mini-International Neuropsychiatric Interview Plus at 12 months | 12 months
  At end of empirical deep brain stimulator programming period
Change from baseline United Parkinsons Disease Rating Scale parts I, II, IV, V at 3 months | 3 months
  At end of first randomised crossover period for Parkinsons disease
Change from baseline United Parkinsons Disease Rating Scale parts I, II, IV, V at 6 months | 6 months
  At end of second randomised crossover period for Parkinsons disease
Change from baseline United Parkinsons Disease Rating Scale parts I, II, IV, V at 12 months | 12 months
  At end of empirical deep brain stimulator programming period for Parkinsons disease
Change from baseline Abnormal Involuntary Movement Scale at 3 months | 3 months
  At end of first randomised crossover period for Parkinsons disease
Change from baseline Abnormal Involuntary Movement Scale at 6 months | 6 months
  At end of second randomised crossover period for Parkinsons disease
Change from baseline Abnormal Involuntary Movement Scale at 12 months | 12 months
  At end of empirical deep brain stimulator programming period for Parkinsons disease

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lind, MBChB, FRACS, Principal Investigator — The University of Western Australia
Locations (1):
- Sir Charles Gairdner Hospital, Perth, Western Australia, Australia